CLINICAL TRIAL: NCT00764855
Title: Validation of the Effect of Propofol and Opiates Closed-loop Administration Device During Anesthesia and Sedation
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/250
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Surgery With General Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients undergoing a surgery with general anesthesia
  Interventions: Procedure: Automatic administration of propofol and opiates during routine clinical practice

INTERVENTIONS:
Procedure: Automatic administration of propofol and opiates during routine clinical practice — The clinical effect of administration of pharmaca can be measured in the changes of heartbeat, blood pressure, respiration and the changes of brain activity by registering EEG. These measurements are performed standard, to secure the safety of the patient.
  The heartbeat and the EEG will be measured by non invasive adhesive electrodes on the skin of the patient.
  The blood pressure will be measured by non invasive blood pressure cuff around the arm and the respiration parameters will be measured by non invasive spirometry, which are all standard available on a anesthesia device.

SUMMARY:
Sleeping medication and analgesia are standard administered during anesthesia. Sleeping medication, Propofol (Diprivan, AstraZeneca), and analgesia, Remifentanil (GlaxoSmithKline), are most frequently used In the University Hospital Ghent.

The clinical effect of administration of pharmaca can be measured in the changes of heartbeat, blood pressure, respiration and the changes of brain activity by registering EEG. These measurements are performed standard, to secure the safety of the patient.

The heartbeat and the EEG will be measured by non invasive adhesive electrodes on the skin of the patient.

The blood pressure will be measured by non invasive blood pressure cuff around the arm and the respiration parameters will be measured by non invasive spirometry, which are all standard available on a anesthesia device.

Most of the pharmaca are administered by a fixed dosage schedule based on the patient's weight.

A more individualized administration of this pharmaca could lead to a better anesthesia quality.

Since considerable time, we know that a computer-controlled administration of these products by automatic coupling between the measured effects and the "spuit"pump to administer the product, could lead to a better administration, optimalisation of the administered dose, because the patients individual effect of the administration can be taken in consideration. This device is called the "closed-loop system". The department of Anesthesia has already proofed the utility of the device for automatic administration of Propofol and opiates in small specific patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a surgery with general anesthesia
* Between 18 and 65 years of age
* Patient signed an informed consent

Exclusion Criteria:

* Patients that did not signed an informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a surgery with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To analyse and to validate the "closed-loop system" of the optimal function of this system for automatic administration of propofol and opiates during routine clinical practice | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Michel Struys, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Neckebroek M, Boldingh JHL, De Smet T, Struys MMRF. Influence of Remifentanil on the Control Performance of the Bispectral Index Controlled Bayesian-Based Closed-Loop System for Propofol Administration. Anesth Analg. 2020 Jun;130(6):1661-1669. doi: 10.1213/ANE.0000000000004208. PMID 31107260
- See also: Website of the University Hospital Ghent — http://www.uzgent.be